CLINICAL TRIAL: NCT06097130
Title: Evaluation of the Effect of Different Nutrients on the Gut Microbiota Composition and Metabolic Activity by Using in Vitro Batch Fermentation and Cellular Models
Brief Title: Batch Fermentation and Microbiome Analysis
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 1920NR
Record Dates: First submitted 2023-03-16; First posted 2023-10-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Microbiome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The correlation between diet and microbiota as well as the effect of microbiota on human health is well established. Studies have shown that people following specific diets have different microbiome profile compared to those following traditional or ordinary diets. In order to screen several food ingredients for their effects on human microbiota composition and metabolic activities, in vitro studies are proposed. Nutrients are added in-vitro in fecal sample, eliminating the need for participants to consume any nutritional product. The batch fermentation in vitro system simulates human colonic microbiota from fecal samples, enabling the complex mixture of microorganisms. This system could serve as a simple model to simulate the diversity as well as the metabolism of human colonic microbiota. We will evaluate the effect on nutrient/s on the age specific microbiome via an in vitro fermentation approach for the 0 to 60 year-old period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant aged from 0 to 60 (based on medical history, physical examination and review of childhood growth chart)
* Written informed consent has been obtained from the parent(s)/legally acceptable representative (LAR) of toddlers and teenagers
* Written informed consent has been obtained for participants aged from 14 years old and above
* Child's parent(s)/legal representative or participant is willing and able to fulfill the requirements of the study protocol.
* Ability to collect their or their infant/child's fecal sample.

Exclusion Criteria:

* The parent(s)/legally acceptable representative (LAR) is not able to provide evidence of parental authority or legal representation.
* Participant following a particular regimen of any type such as vegan, vegetarian, ketogenic, paleo diet,
* Chronic or recurrent diarrhea with spontaneous bowel movements more often than 2 times daily,
* Antibacterial/antifungal therapy during the 3 months prior to study enrolment,
* Medications or supplements that are known to alter gut function or microbiota (i.e. acid antisecretory drugs, pre-/probiotics supplements, laxatives) during the 4 weeks prior to study enrolment,
* Prior gastrointestinal surgery (apart from appendectomy, cholecystectomy or herniotomy),
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer,
* Artificially sweetened beverage intake higher than 1000 ml/ per day,
* Current or history of gastrointestinal diseases like (Celiac Disease, Crohn's Disease, Ulcerative colitis, Irritable Bowel Syndrome, infantile colic, recurrent abdominal pain, functional constipation, ulcers, infections (based on anamnesis),
* Participants participating in another interventional study,
* Participants/parents having a hierarchical or family link with the research team members.

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy population
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition | Through study completion, an average of 1 year
  Measured by 16s rRNA sequencing or next Generation Sequencing (NGS) or by qPCR

SECONDARY OUTCOMES:
Change in Short Chain Fatty Acids (SCFA) | Through study completion, an average of 1 year
  Measured using Gas Chromatography (GC)
Change in metabolic profile | Through study completion, an average of 1 year
  Measured using Gas Chromatography (GC) or Gas chromatography-mass spectrometry (GC-MS)
Protein expression of epithelial cells | Through study completion, an average of 1 year
  Measured by western blot

CONTACTS AND LOCATIONS:
Locations (1):
- Nestle Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No